CLINICAL TRIAL: NCT04801004
Title: A Real-world Study to Evaluate the Primary Patency and Freedom From TLR of Endovascular Treatment in TOSAKA III In-stent Restenosis of Lower Extremity Femoropopliteal Artery.
Acronym: FP-Restore
Status: Active, not recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: RenJi Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); Chengdu University of Traditional Chinese Medicine (Other); Xuanwu Hospital, Beijing (Other); First People's Hospital of Hangzhou (Other); Qingdao Hiser Medical Group (Other); Second Affiliated Hospital of Soochow University (Other); Liyuan Hospital of Tongji Medical College of Huazhong University of Science and Technology (Unknown)
Responsible Party: Sponsor
Other Study IDs: The FP-artery Restore study
Record Dates: First submitted 2021-03-10; First posted 2021-03-16 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Arterial Disease
Keywords: in-stent restenosis
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study is a prospective, multi-center, real world, observational study, which aims at evaluating the safety, efficacy and economic cost of endovascular treatments for endovascular therapies in tosaka III (totally occluded) in-stent restenosis.It is estimated that 300 subjects diagnosed with tosaka III in-stent restenosis and receive endovascular treatments will be enrolled in nine centers from April 2021 to December 2022 nation-widely. All the subjects will be under follow-up for 24 months. There is no restriction on the endovascular techniques. The primary outcomes include clinical-driven freedom from TLR at 24 months.

DETAILED DESCRIPTION:
In-stent restenosis was a series of complications of treatment in peripheral artery disease, which lead the fluid of lower extremity re-limited even chronic limb ischemia and amputation. Its typical symptoms were recurrent claudication, rest pain and ischemic. Tosaka III in-stent restenosis, which also called in-stent occlusion was one of the most serious of this kind of complications. Its symptoms usually more severe and irreversible, and its treatments were complicated and challenging. The efficacy of single balloon angioplasty is limited. New devices including drug-coated balloon, intravascular Lithotripsy, directional atherectomy, laser debulking devices and stent-grafts offer another chance and better prognosis. The data of these new devices, however, are mainly from low-quality evidence. Therefore, we start this prospective, multicenter, real-world, observational study, providing new data on the safety, efficacy and health economics evaluation of endovascular treatments for Tosaka III in-stent restenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Tosaka III In-stent restenosis after stent implantation in PAD patients (Including acute and subacute thrombotic lesions).
2. Rutherford grade 2-5.
3. Stents should be located in the femoropopliteal artery.
4. The stenosis of iliac artery on the affected side is less than 30% or the residual stenosis after treatment is less than 30%.
5. Informed consent has been signed

Exclusion Criteria:

1. Tosaka I or II in-stent restenosis.
2. Stents are located in iliac artery or artery below the knee, or the preoperative CTA showed type 3 or 4 stent fracture.
3. Rutherford Grade 6.
4. Thromboangiitis obliterans (TAO)-based, arteritis-based or connective tissue disorder-based FP-ISR.
5. Intraoperative conversion to hybrid or open surgery.
6. Patients refusing to sign informed consent forms.
7. Life expectancy of patients is less than 12 months.
8. The pregnant or nursing patients.
9. The patients with severe ischemia of lower extremity who would receive major amputation in plan.
10. Patients in whom antiplatelet or anticoagulant therapy is contraindicated.
11. Myocardial infarction or stroke within 3 months prior to enrolment.
12. Patient with known allergy to contrast agents or medications used to perform endovascular intervention.
13. Patients participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the primary endpoint.
14. Patients who refuse to cooperate with long-term follow-up or who have difficulty communicating.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients with Tosaka III in-stent restenosis lower extremity femoropopliteal artery.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from clinically-driven TLR | 24 months
  CD-TLR was deﬁned as any reintervention within the target lesion(s) because of recurrent symptoms. Freedom form CD-TLR were defined as the rates of the number of patients who did not receive reintervention verse the number of patients during the follow-up period.

SECONDARY OUTCOMES:
Primary patency | 1month, 6 months,12 months, 18 months ,24 months
  The primary patency rate was defined as the percentage of stent patency examined by DUS or CTA examination of lower limb arteries during follow-up.
Technical success rate | 30 days
  Successfully revascularize the target vessel. The residual stenosis is <30% and there is no acute thrombosis occurred in the target vessel within 30 days post-operation. The Technical success rate was defined as the rate of the number of patients who receive the treatment as intended verse the number of the patients enrolled.
Incidence of major adverse events. | 1month, 3 months,6 months, 12 months ,24 months
  Major adverse events include anyone of the following: all-cause mortality, Myocardial infarction, ischemic stroke, acute limb ischemia, and major amputation of a vascular etiology, and arterial thrombosis related to endovascular manipulation.
Freedom from TLR | 1month, 6 months,12 months, 18 months
  TLR was deﬁned as a reintervention performed for >50% diameter stenosis or in the target lesion after documentation of recurrent clinical symptoms following the index procedure or bailout stenting during the index procedure. Freedom form TLR were defined as the rates of the number of patients who did not receive reintervention verse the number of patients during the follow-up period.
Vascular quality of life questionnaire(VascuQol) | 3 months,6 months, 12 months ,24 months
  The VascuQol was designed as a questionnaire containing five domains: pain (4 items), symptoms (4 items), activities (8 items), social (2 items), and emotional (7 items) to evaluate Health related quality of life (HRQL). Every item has seven response options, with scores ranging from 1 to 7. A total score is the sum of all 25 item scores divided by 25.And both the total score as well as the domain scores range from 1 (worst HRQL) to 7 (best HRQL).The lower the value, the poorer the quality of life.
Health economics evaluation | 24months
  All the cost related to the target vessel and spent in the inpatient ward will be recorded and analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China

REFERENCES:
- [Background] Tosaka A, Soga Y, Iida O, Ishihara T, Hirano K, Suzuki K, Yokoi H, Nanto S, Nobuyoshi M. Classification and clinical impact of restenosis after femoropopliteal stenting. J Am Coll Cardiol. 2012 Jan 3;59(1):16-23. doi: 10.1016/j.jacc.2011.09.036. PMID 22192663
- [Background] Armstrong EJ, Thiruvoipati T, Tanganyika K, Singh GD, Laird JR. Laser Atherectomy for Treatment of Femoropopliteal In-Stent Restenosis. J Endovasc Ther. 2015 Aug;22(4):506-13. doi: 10.1177/1526602815592133. Epub 2015 Jun 30. PMID 26130385
- [Background] Dippel EJ, Makam P, Kovach R, George JC, Patlola R, Metzger DC, Mena-Hurtado C, Beasley R, Soukas P, Colon-Hernandez PJ, Stark MA, Walker C; EXCITE ISR Investigators. Randomized controlled study of excimer laser atherectomy for treatment of femoropopliteal in-stent restenosis: initial results from the EXCITE ISR trial (EXCImer Laser Randomized Controlled Study for Treatment of FemoropopliTEal In-Stent Restenosis). JACC Cardiovasc Interv. 2015 Jan;8(1 Pt A):92-101. doi: 10.1016/j.jcin.2014.09.009. Epub 2014 Dec 10. PMID 25499305
- [Background] Kokkinidis DG, Behan S, Jawaid O, Hossain P, Giannopoulos S, Singh GD, Laird JR, Valle JA, Waldo SW, Armstrong EJ. Laser atherectomy and drug-coated balloons for the treatment of femoropopliteal in-stent restenosis: 2-Year outcomes. Catheter Cardiovasc Interv. 2020 Feb 15;95(3):439-446. doi: 10.1002/ccd.28636. Epub 2019 Dec 9. PMID 31816169
- [Background] Li X, Zhou M, Ding Y, Wang Y, Cai L, Shi Z. A systematic review and meta-analysis of the efficacy of debulking devices for in-stent restenosis of the femoropopliteal artery. J Vasc Surg. 2020 Jul;72(1):356-366.e5. doi: 10.1016/j.jvs.2019.11.058. Epub 2020 Feb 21. PMID 32093910
- [Background] Kinstner CM, Lammer J, Willfort-Ehringer A, Matzek W, Gschwandtner M, Javor D, Funovics M, Schoder M, Koppensteiner R, Loewe C, Ristl R, Wolf F. Paclitaxel-Eluting Balloon Versus Standard Balloon Angioplasty in In-Stent Restenosis of the Superficial Femoral and Proximal Popliteal Artery: 1-Year Results of the PACUBA Trial. JACC Cardiovasc Interv. 2016 Jul 11;9(13):1386-92. doi: 10.1016/j.jcin.2016.04.012. PMID 27388828
- [Background] Bosiers M, Deloose K, Callaert J, Verbist J, Hendriks J, Lauwers P, Schroe H, Lansink W, Scheinert D, Schmidt A, Zeller T, Beschorner U, Noory E, Torsello G, Austermann M, Wauters J. Stent-grafts are the best way to treat complex in-stent restenosis lesions in the superficial femoral artery: 24-month results from a multicenter randomized trial. J Cardiovasc Surg (Torino). 2020 Oct;61(5):617-625. doi: 10.23736/S0021-9509.20.11382-X. PMID 33231029
- [Background] Shammas NW, Petruzzi N, Henao S, Armstrong EJ, Shimshak T, Banerjee S, Latif F, Eaves B, Brothers T, Golzar J, Shammas GA, Jones-Miller S, Christensen L, Shammas WJ. JetStream Atherectomy for the Treatment of In-Stent Restenosis of the Femoropopliteal Segment: One-Year Results of the JET-ISR Study. J Endovasc Ther. 2021 Feb;28(1):107-116. doi: 10.1177/1526602820951916. Epub 2020 Sep 4. PMID 32885736
- [Background] Torsello G, Stavroulakis K, Brodmann M, Micari A, Tepe G, Veroux P, Benko A, Choi D, Vermassen FEG, Jaff MR, Guo J, Dobranszki R, Zeller T; IN.PACT Global Investigators. Three-Year Sustained Clinical Efficacy of Drug-Coated Balloon Angioplasty in a Real-World Femoropopliteal Cohort. J Endovasc Ther. 2020 Oct;27(5):693-705. doi: 10.1177/1526602820931477. Epub 2020 Jun 25. PMID 32583749
- [Background] Tepe G, Schroeder H, Albrecht T, Reimer P, Diehm N, Baeriswyl JL, Brechtel K, Speck U, Zeller T. Paclitaxel-Coated Balloon vs Uncoated Balloon Angioplasty for Treatment of In-Stent Restenosis in the Superficial Femoral and Popliteal Arteries: The COPA CABANA Trial. J Endovasc Ther. 2020 Apr;27(2):276-286. doi: 10.1177/1526602820907917. Epub 2020 Feb 25. PMID 32096451
- [Derived] Li X, Zhou M, Ding Y, Wu Z, Feng Z, Guo L, Li Q, Fang X, Sang H, Ye M, Shi Z. Design of the FP-RESTORE study: a protocol for prospective, observational study of real-world treatments with endovascular therapy in patients with femoropopliteal artery Tosaka III in-stent restenosis. BMJ Open. 2022 Dec 6;12(12):e060200. doi: 10.1136/bmjopen-2021-060200. PMID 36600357